CLINICAL TRIAL: NCT00746083
Title: Randomized Controlled Trial for Health Promotion/ Obesity Prevention Targeting Low-income, Urban, African-American Adolescents
Brief Title: Challenge!, a Health Promotion/ Obesity Prevention Program for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Annie E. Casey Foundation (Other Government); The Thomas Wilson Sanitarium for Children of Baltimore City (Other); Johns Hopkins Bloomberg School of Public Health (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Maureen Black, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-21033; R40MC00241, M01 RR16500
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Overweight
Keywords: pediatric; obesity; African American; adolescents; intervention; home-based; community-based
MeSH Terms: conditions — Overweight; Obesity | interventions — Human Challenge Trials as Topic; Organizational Objectives; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Challenge!
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Challenge! — Each adolescent in the intervention group received 12 lessons administered in adolescent's home or community by a "personal trainer" (a college-aged mentor). The lessons focused on behavior change relating to diet and physical activity and was based on social cognitive theory. At the end of each lesson the adolescent set a behavior change goal for themselves. The adolescents were taught how to track their goals and they discussed thir ability/inability to meet their goals at each meeting with their personal trainer.
  Other Names: Obesity prevention; Goal setting; Diet; Physical activity
  Arms: Intervention group

SUMMARY:
The purpose of Challenge! is to determine if adolescents enrolled in a health promotion/ obesity prevention program will have a healthier BMI-for-age z-score and body composition (body fat %), will consume a healthier diet, and engage in higher levels of physical activity compared to those that did not receive the intervention over time.

DETAILED DESCRIPTION:
Pediatric overweight is a major public health problem in the US, with the prevalence of overweight among children of all ages increasing dramatically over the past several decades. Interventions aimed at reducing the increased weight gain during adolescence have produced mixed results.

Challenge! is a randomized controlled trial for health promotion/ obesity prevention targeting low-income, urban, African American adolescents. Healthy adolescents were recruited from an urban medical center and from local middle schools. Weight status was not part of the inclusion criteria.

The intervention was home- and community-based and delivered one-on-one to each adolescent by a college-age "personal trainer". The intervention focused on goal-setting, consuming a healthy diet (increase fruits, vegetables, and water, and decrease high-fat snack and convenience foods), and increasing physical activity. We hypothesized that the teens enrolled in the intervention would have a healthier BMI-for-age z-score and a healthier body composition (body fat %) compared to those that did not receive the intervention over time. Additionally, we hypothesized that those enrolled in the intervention would consume healthier diets and have higher levels of physical activity compared to those that did not receive the intervention over time.

ELIGIBILITY:
Inclusion Criteria:

* Ages 11-16, willing to participate in a randomized controlled trial for health promotion

Exclusion Criteria:

* Outside of age range

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2001-04; Primary Completion 2005-07 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
BMI-for-age z-score and percentiles (measured weight and height, self-reported gender and date of birth)and Body composition (Dual Energy X-ray Absorptiometry, and Bioelectrical Impedance Analysis) | 2 years

SECONDARY OUTCOMES:
Physical Activity (accelerometry and self-report) Diet (Food frequency questionnaire) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M Black, PhD, Principal Investigator — University of Maryland School of Medicine, Department of Pediatrics, United States
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Snitker S, Le KY, Hager E, Caballero B, Black MM. Association of physical activity and body composition with insulin sensitivity in a community sample of adolescents. Arch Pediatr Adolesc Med. 2007 Jul;161(7):677-83. doi: 10.1001/archpedi.161.7.677. PMID 17606831
- [Background] Mitola AL, Papas MA, Le K, Fusillo L, Black MM. Agreement with satisfaction in adolescent body size between female caregivers and teens from a low-income African-American community. J Pediatr Psychol. 2007 Jan-Feb;32(1):42-51. doi: 10.1093/jpepsy/jsl004. Epub 2006 Jun 8. PMID 16762992
- [Derived] Devonshire AL, Hager ER, Black MM, Diener-West M, Tilton N, Snitker S. Elevated blood pressure in adolescent girls: correlation to body size and composition. BMC Public Health. 2016 Jan 26;16:78. doi: 10.1186/s12889-016-2717-6. PMID 26812968
- [Derived] Black MM, Hager ER, Le K, Anliker J, Arteaga SS, Diclemente C, Gittelsohn J, Magder L, Papas M, Snitker S, Treuth MS, Wang Y. Challenge! Health promotion/obesity prevention mentorship model among urban, black adolescents. Pediatrics. 2010 Aug;126(2):280-8. doi: 10.1542/peds.2009-1832. Epub 2010 Jul 26. PMID 20660556